CLINICAL TRIAL: NCT04402255
Title: The Effect of Pilates Based Exercise Practice on Physical and Psychological Parameters in Patients With Behçet and Familial Mediterranean Fever.
Brief Title: Pilates Based Exercises in Patients With Behçet and Familial Mediterranean Fever.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nejla Uzun, MSc, Pt, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83088843-604.01.04-5578
Record Dates: First submitted 2020-05-17; First posted 2020-05-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2020-05

CONDITIONS: Behcet Disease; FMF
MeSH Terms: conditions — Behcet Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- behcet group (Experimental): this group includes 16 patients with behçet
  Interventions: Other: pilates exercise
- fmf group (Experimental): this group includes 16 patients with fmf
  Interventions: Other: pilates exercise
- healty control (Active Comparator): this group includes 16 healthy control
  Interventions: Other: pilates exercise

INTERVENTIONS:
Other: pilates exercise — The key elements of Pilates during supine, prone, side-lying and standing positions will be taught. These key elements are: breathing (diaphragmatic), focusing (neutral position), rib cage placement, shoulder placement, head and neck placement (neutral position). Then, Pilates based 'mat' exercises will be performed by the physiotherapist in the clinic for 8 weeks, 2 days / week, 16 sessions. Each session will be programmed to be 45 minutes. During all exercises, including warm-up and cooling, patients will be asked to provide key elements and protect them during movements. Depending on the condition of the patients, the exercises will be advanced from easy to difficult.

SUMMARY:
Behcet's disease (BD) is a chronic systemic inflammatory disease which is characterized by oral and genital ulcers, uveitis and skin lesions. Musculoskeletal involvement such as arthritis, arthralgia, enthesitis and sacroiliitis can be seen in the course of BD. Familial Mediterranean fever (FMF) is the most frequent autoinflammatory disease (AID) and characterized by selflimited episodes of fever and polyserositis. It is the most common monogenic periodic fever syndrome that affects mainly the people of Mediterranean descent. Regular physical activity involving aerobic and strengthening programs in inflammatory rheumatic diseases has a long-term anti-inflammatory effect. Eccentric exercises cause an acute increase in TNF alpha level and should be avoided especially at the beginning. It has been stated that patients should be encouraged about aerobic exercise programs where the intensity is gradually increased, starting with low intensity. Pilates method is the mind and body centering technique developed by Joseph Hubertus Pilates, based on providing lumbopelvic stability. FMF and BH have common characteristics such as ethnicity, etiopathogenetic mechanisms, symptoms, and treatment. When we look at the literature, there is no study on the effectiveness of exercise applications in FMF and Behçet patients. The purpose of our study; It is the comparison of the effectiveness of physical activity in patients diagnosed with Behçet and FMF and healthy individuals. In this context, with the short form of the International Physical Activity Evaluation Questionnaire, Behçet's patients whose physical activity level is inactive will be Group 1, FMF patients Group 2 and healthy controls with similar demographic characteristics will be Group 3. Pilates based exercise program will be applied to all 3 groups for 8 weeks, 2 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Being inactive or minimally active according to the International Physical Activity Survey
* Being between the ages of 18-65
* Being diagnosed with FMF at least 1 year ago according to diagnostic criteria
* A diagnosis of BH at least 1 year ago according to the International Behçet Working Group
* Having a cooperative level that can adapt to the evaluation and exercise program

Exclusion Criteria:

* Those with any central nervous system involvement that may interfere with exercise
* Those who do not want to participate in the study
* Pregnant women
* Having other chronic diseases
* Psychiatric disorders and treated
* Those with cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) Web sonuçları International Physical Activity Questionnaire - Short Form | change from baseline to 8 weeks, follow up at two months
  The BBS is a 14- item balance test recognized as the gold standard tool for assessing balance (higher scores indicate better balance)
six minute walk test | change from baseline to 8 weeks, follow up at two months
  It is a simple test that measures the distance an individual can walk at a fast pace on a flat, hard floor in 6 minutes.
Biodex balance system (BBS) | change from baseline to 8 weeks, follow up at two months
  The BBS has a round foot platform that moves in all planes. It grants 20 degrees of foot platform motion in different directions. The platform has foot angles and heel coordinates for proper foot placement before starting the balance test trial. The foot angles range from 0° to 45° and heel coordinates are expressed as the intersection of letters from A to P and numbers from 1 to 21. The participants were asked to centralize their body while they placed their feet in the most comfortable position and their feet 10 cm apart with eyes open. They were asked to hold the rails in case they felt unbalanced. The machine measured the magnitude of their postural sways: higher scores for postural sway indicate impaired balance, and a lower score indicate excellent balance

SECONDARY OUTCOMES:
international physical activity questionnaire- short form | change from baseline to 8 weeks, follow up at two months
  This short questionnaire, consisting of seven questions, evaluates the amount of walking done in the last week and the amount of moderate and difficult physical activities performed in work, transportation, housework, gardening and leisure activities.
Hamilton Depression Scale | change from baseline to 8 weeks, follow up at two months
  The scale was prepared as 21 items, but the last four items were not included in the scoring. The total score is determined on 17 items.
Nottingham Health Profile Questionnaire (NHP) | change from baseline to 8 weeks, follow up at two months
  NHP were used as research tools. The Nottingham Health Profile Questionnaire was used to measure health problems perceived by the patient and to assess the effect of these problems on daily functioning

CONTACTS AND LOCATIONS:
Locations (1):
- IstanbulU, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No